CLINICAL TRIAL: NCT00539344
Title: A Phase 1, Open-Label, Dose Escalation Study of ANG1005 in Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angiochem Inc (Industry)
Responsible Party: Jean-Paul Castaigne, MD - President & CEO, Angiochem Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ANG1005-CLN-01; FDA
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Recurrent or Progressive Malignant Glioma
Keywords: Glioblastoma multiforme; Anaplastic astrocytoma; Anaplastic oligodendroglioma
MeSH Terms: conditions — Recurrence; Glioblastoma; Astrocytoma; Oligodendroglioma | interventions — paclitaxel-Angiopep-2 conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ANG1005

INTERVENTIONS:
Drug: ANG1005 — IV infusion once every 21 days

SUMMARY:
This is a phase 1, multi-centre, sequential cohort, open-label, dose-escalation study of the safety, tolerability, and PK of ANG1005 in patients with recurrent or progressive malignant glioma. ANG1005 will be given by IV infusion once every 21 days (1 treatment cycle). Each patient will participate in only 1 dose group and will receive up to 6 cycles of treatment provided there is no evidence of tumor progression, there is recovery to ≤Grade 1 or baseline nonhematologic, ANG1005-related toxicity (except alopecia), the absolute neutrophil count is ≥1.5 x 109/L, and the platelet count is ≥100 x 109/L.

DETAILED DESCRIPTION:
This is a phase 1, multi-centre, sequential cohort, open-label, dose-escalation study of the safety, tolerability, and PK of ANG1005 in patients with recurrent or progressive malignant glioma. ANG1005 will be given by IV infusion once every 21 days (1 treatment cycle). Each patient will participate in only 1 dose group and will receive up to 6 cycles. Patients may receive additional cycles of ANG1005 if there is no evidence of tumor progression, there is recovery to ≤Grade 1 or baseline nonhematologic, ANG1005-related toxicity (except alopecia), the absolute neutrophil count is ≥1.5 x 109/L, and the platelet count is ≥100 x 109/L.

Initially, cohorts of 1 - 3 patients will be enrolled into each dose group. Dose escalation by dose doubling will be done for the first 3 dose groups followed by a modified Fibonacci dose escalation scheme with increases of 67%, 50%, 40% and 33% thereafter. If > 1 patient in a cohort experience an emergent ≥ Grade 2 drug-related toxicity during the first treatment cycle, then a minimum of 3 patients will be enrolled into that, and all subsequent cohort(s) and dose doubling will be stopped if applicable.

If > 1 patient in a cohort experience a dose limiting toxicity (DLT) during the first treatment cycle, defined as any of the following that are both treatment-emergent and at least possibly related to ANG1005: i) Any Grade 3 or 4 nonhematologic toxicity, ii) Febrile neutropenia, iii) Grade 4 neutropenia of ≥7 days duration, and/or iv) Any Grade 4 thrombocytopenia, then dose escalation will stop and prior doses will be explored as the maximum tolerated dose (MTD), that dose-level at which ≤1 of 6 patients in a cohort develop an emergent DLT).

Once the MTD is established, approximately 14 patients will be enrolled at that dose-level in order to further assess the safety and tolerability of ANG1005, the PK profile of ANG1005 at the MTD, and the preliminary anti-tumor activity of ANG1005 in patients with malignant glioma.

Approximately 8 additional patients who are scheduled for debulking surgery for recurrent disease may be enrolled into a separate sub-study to obtain preliminary information about whether or not ANG1005 crosses the blood-brain barrier into malignant glioma tumors. These patients will receive ANG1005 prior to surgery at the dose level established to be safe and tolerable at that time and may continue to receive additional cycles of ANG1005 following surgery, if appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Histologically confirmed malignant glioma
3. Radiologically confirmed progression of malignant glioma
4. Patients must, in the opinion of the investigator, be ineligible for current standard of care treatment
5. No evidence of acute intracranial/intratumoral hemorrhage
6. Male and female patients
7. Age ≥18 years
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
9. An expected survival of at least 3 months
10. Measurable disease according to Macdonald response criteria
11. Male and female subjects who are not surgically sterile or post-menopausal must agree to use reliable methods of birth control for the duration of the study and for 90 days after the last dose of study drug administration; male partners of female subjects should use condoms for the duration of the study, and for 90 days after the last dose of study drug administration

Exclusion Criteria:

1. Chemotherapy, radiotherapy (except palliative radiation delivered to <20% of bone marrow), or investigational agents within 4 weeks before the first dose of study drug. Biologic therapy (such as 13-cis-retinoic acid, thalidomide, tamoxifen, celebrex, erlotinib, imatinib, vorinostat, and lapatinib) and immunotherapy (such as interferon a or b, cdx-110 (EGFR vIII vaccine), interleukin 2, thalidomide) within 1 week before the first dose of study drug. Bevacizumab within 6 weeks before the first dose of study drug
2. Pregnant or lactating females
3. Any acute viral, bacterial, or fungal infection that requires parenteral therapy within 14 days prior to study treatment
4. Known severe hypersensitivity to paclitaxel
5. Severe toxicity with previous taxane treatment
6. Patients being treated with P450 CYP 3A4 or CYP 2C8 enzyme-inducing anti-convulsant drugs within 14 days prior to treatment with study drug
7. Patients with inadequate hematological, liver, and renal function
8. Known or suspected acute or chronic active Hepatitis B, or Hepatitis C or HIV/AIDS
9. Patients with unstable or uncompensated respiratory, cardiac, hepatic or renal disease or any other organ system dysfunction, medical condition, or laboratory abnormality which, in the opinion of the investigator, would either comprise the patient's safety or interfere with the evaluation of the test material
10. Evidence of persistent Grade 2 or greater neurotoxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of intravenously administered ANG1005 in patients with malignant glioma. | On-going
To identify the maximum tolerated dose (MTD) of ANG1005 in patients with malignant glioma. | End of dose escalation

SECONDARY OUTCOMES:
To examine the pharmacokinetics (PK) of ANG1005. | End of study
To confirm the safety and tolerability of ANG1005 at the MTD. | End of dose escalation
To assess the immunogenicity of ANG1005. | End of study
To obtain preliminary information about the antitumor activity of ANG1005 in patients with malignant glioma. | On-going
To obtain preliminary information about whether or not ANG1005 crosses the blood- brain barrier into malignant glioma tumors (Sub-study). | On-going

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Irving Comprehensive Cancer Center, Columbia University Medical Center, New York, New York
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - UT Health Science Center at the Cancer Therapy and Research Center (CTRC), San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Result] Drappatz J, Brenner A, Wong ET, Eichler A, Schiff D, Groves MD, Mikkelsen T, Rosenfeld S, Sarantopoulos J, Meyers CA, Fielding RM, Elian K, Wang X, Lawrence B, Shing M, Kelsey S, Castaigne JP, Wen PY. Phase I study of GRN1005 in recurrent malignant glioma. Clin Cancer Res. 2013 Mar 15;19(6):1567-76. doi: 10.1158/1078-0432.CCR-12-2481. Epub 2013 Jan 24. PMID 23349317
- See also: Related Info — http://www.angiochem.com